CLINICAL TRIAL: NCT02046525
Title: Restoration of the Fecal Microbiome After Antimicrobial Exposure With Autologous Fecal Flora Restoration Therapy
Brief Title: Autologous Fecal Therapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 201312022; 1U54CK000162 (NIH)
Record Dates: First submitted 2014-01-23; First posted 2014-01-27 (Estimated); Results first posted 2019-05-22 (Actual); Last update posted 2019-06-04 (Actual); Status verified 2019-05

CONDITIONS: Infectious Disease of Digestive Tract
Keywords: Fecal microbiota therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Auto fecal microbitoa therapy (Experimental): autologous fecal microbiota therapy
  Interventions: Biological: Autologous fecal microbiota therapy
- Saline enema (Placebo Comparator): Saline enema
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: Autologous fecal microbiota therapy
  Arms: Auto fecal microbitoa therapy
Other: Placebo — Saline enema
  Arms: Saline enema

SUMMARY:
Ten healthy volunteers will be recruited to receive either an autologous stool transplant or a saline enema to determine if autologous fecal microbiota therapy will be able to rapidly, and safely, restore a patient's fecal microbiome after antimicrobial exposure.

ELIGIBILITY:
Inclusion Criteria:

Healthy Adults 18-70 years of age-

Exclusion Criteria:

history of allergic reaction to beta-lactam antimicrobials; any non-topical antimicrobial exposure or tube feeds as a primary source of nutrition in the past six months; pregnant or risk of becoming pregnant during the study period; gastroenteritis in the last 3 months; incontinent of stool; prior resection or alteration of the stomach; small bowel, or colon; unwillingness to receive an enema/FMT; known colonization with an MDRO; anticipated change in diet or medications, or elective surgery, during the study period; or a history of an intestinal disorder -

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2014-03; Primary Completion 2018-12 (Actual); Study Completion 2018-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Washington University in St. Louis, St Louis, Missouri, United States

REFERENCES:
- [Derived] Bulow C, Langdon A, Hink T, Wallace M, Reske KA, Patel S, Sun X, Seiler S, Jones S, Kwon JH, Burnham CA, Dantas G, Dubberke ER. Impact of Amoxicillin-Clavulanate followed by Autologous Fecal Microbiota Transplantation on Fecal Microbiome Structure and Metabolic Potential. mSphere. 2018 Nov 21;3(6):e00588-18. doi: 10.1128/mSphereDirect.00588-18. PMID 30463925

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Auto Fecal Microbitoa Therapy | Saline Enema
Started | 5 | 5
Completed | 5 | 5
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Auto Fecal Microbitoa Therapy | Saline Enema | Total
Number analyzed (Participants) | 5 | 5 | 10
Age, Continuous [Median (Full Range); unit: years] | 26 [25 to 57] | 34 [24 to 56] | 31 [24 to 57]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 2 | 6
  Male | 1 | 3 | 4
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Non-white race | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 5 | 5 | 10

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Restoration of Microbial Community Composition to the Pre-antibiotic State by 90 Days Post FMT or Saline Enema
Description: Restoration of microbial community composition (bacterial taxa that are present) and structure (abundance of taxa) to the subject's state prior to antimicrobial exposure. Bacterial taxa are the types/strains of bacteria found in the microbiome.
Time Frame: 90 days after enrollment
Measure: Count of Participants; unit: Participants
Groups:
- Auto Fecal Microbiota Therapy: autologous fecal microbiota therapy
  Autologous fecal microbiota therapy
Arm/Group | Auto Fecal Microbiota Therapy | Saline Enema
Number analyzed (Participants) | 5 | 5
Participants | 5 | 5

ADVERSE EVENTS:
Time Frame: 90 days post-enema
Arm/Group | Auto Fecal Microbitoa Therapy | Saline Enema
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/5
Other Adverse Events (participants affected / at risk) | 1/5 | 1/5
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Auto Fecal Microbitoa Therapy (N=5) | Saline Enema (N=5)
Ear infection (Infections and infestations) | 0 (0) | 1 (1)
H. pylori infection (Infections and infestations) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-12-11): https://cdn.clinicaltrials.gov/large-docs/25/NCT02046525/Prot_SAP_000.pdf